CLINICAL TRIAL: NCT05441410
Title: Comparing Safety and Protective Efficacy of the Whole Plasmodium Falciparum Sporozoite Chemoprophylaxis Vaccine Candidate PfSPZ-CVac and Prime- Target Vaccination with Viral Vectored Vaccine Candidate Regime MVA ME-TRAP/ ChAd63 ME-TRAP in Malaria-naïve, Healthy Adult Volunteers in Germany
Brief Title: Comparing Safety and Protective Efficacy of Vaccine Candidate PfSPZ-CVac and MVA ME-TRAP/ ChAd63 ME-TRAP in Adults
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Sanaria Inc. (Industry); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPICY
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: There will be two groups: Group 1 ("PfSPZ-CVac") and Group 2 ("ME-TRAP"). Within Group 1, Arm 1 (N=12) participants will receive PfSPZ Challenge (NF54) via direct venous inoculation (DVI) along with one weight-adjusted oral dose of Pyramax on day 1, day 6, and day 29. The placebo group of Arm 2 (N=3) will receive an oral placebo pill and saline DVI on day 1, day 6, and day 29.
  In Group 2, participants of Arm 1 (N=12) will receive MVA ME-TRAP intramuscularly on day 1 and ChAd63 ME-TRAP intravenously by DVI on day 29. The placebo group of Arm 2 (N=3) will receive saline intramuscularly on day 1 and intravenously on day 29.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PfSPZ-CVac/Pyramax (Experimental): 200.000 PfSPZ of PfSPZ Challenge NF54 will be administered by DVI along with one weight-adjusted oral dose of Pyramax each on day 1, day 6, and day 29
  Interventions: Drug: Pyronaridine Tetraphosphate, Artesunate Drug Combination; Biological: PfSPZ Challenge (NF54)
- MVA ME-TRAP/ChAd63 ME-TRAP (Experimental): MVA ME-TRAP 1.5 x 10^8 pfu will be administered intramuscularly on day 1 for priming. ChAd63 ME-TRAP 5 x 10^10 vp will subsequently administered by DVI on day 29.
  Interventions: Biological: MVA ME-TRAP; Biological: ChAd63 ME-TRAP
- Saline/placebo pill (Placebo Comparator): As placebo comparator to PfSPZ-CVac/Pyramax, saline will be administered intravenously along with an oral placebo pill on day 1, day 6, and day 29.
  As placebo comparator to MVA ME-TRAP/ChAd63 ME-TRAP, saline will be administered intramuscularly on day 1 and intravenously on day 29. No placebo pill will be used to compare to the arm MVA ME-TRAP/ChAd63 ME-TRAP.
  Interventions: Biological: Sodium chloride (NaCl) 0.9%

INTERVENTIONS:
Drug: Pyronaridine Tetraphosphate, Artesunate Drug Combination — Combination drug for treatment of uncomplicated malaria
  Other Names: Pyramax
  Arms: PfSPZ-CVac/Pyramax
Biological: PfSPZ Challenge (NF54) — cryopreserved Plasmodium falciparum sporozoites injected by intravenous inoculation
  Arms: PfSPZ-CVac/Pyramax
Biological: MVA ME-TRAP — virally vectored subunit vaccine candidates where ME-TRAP is expressed by the non-replicating viral vector Modified Vaccinia Ankara (MVA)
  Arms: MVA ME-TRAP/ChAd63 ME-TRAP
Biological: ChAd63 ME-TRAP — virally vectored subunit vaccine candidates where ME-TRAP is expressed by the non-replicating viral vector Chimpanzee Adenovirus 63 (ChAd63)
  Arms: MVA ME-TRAP/ChAd63 ME-TRAP
Biological: Sodium chloride (NaCl) 0.9% — 0.9% NaCl solution for injection
  Other Names: Placebo: Saline
  Arms: Saline/placebo pill

SUMMARY:
This is a single centre, randomized, placebo-controlled phase 1/2 study comparing two malaria vaccine candidates. The first vaccine candidate PfSPZ-CVac (Plasmodium falciparum sporozoites (PfSPZ) challenge administered with a chemoprophylactic antimalarial) will be chemoattenuated in vivo with the antimalarial Pyramax. The second vaccine candidate is prime- target vaccination with viral vectored vaccine candidate regime MVA ME-TRAP (Modified Vaccinia Ankara (MVA) multiple epitope thrombosponin-related adhesion protein (ME-TRAP)) and ChAd63 ME-TRAP (Chimpanzee adenovirus 63 (ChAd63). The safety and protective efficacy of both vaccine candidates will be to assessed by controlled human malaria infection with PfSPZ Challenge strain NF54 administered intravenously by syringe.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner if required.
* Residence in Tübingen or surroundings for the period of the trial.
* Women only: Must agree to practice continuous highly effective contraception for the duration of the study and until the end of relevant systemic exposure (a method which results in a low failure rate; i.e. less than 1% per year). Additionally, women will only be exposed to the PfSPZ-CVac/ME-TRAP products following a negative highly sensitive pregnancy test the day before immunization/CHMI.
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local and national blood banking eligibility criteria (which is a permanent refrain from blood donations after a malaria parasite infection).
* Provision of written informed consent to receive PfSPZ Challenge products or ME-TRAP products for immunization and subsequently for CHMI.
* Accept to be contacted (24/7) by mobile phone during the immunization and CHMI period.
* Willingness to take Pyramax during immunization (PfSPZ-CVac group) and a curative antimalarial regimen following CHMI.
* Agreement to stay overnight for observation during the period of intensive follow-up post-challenge if required.
* Answer all questions on the informed consent quiz correctly.
* A body mass index <35

Exclusion Criteria:

* History of P. falciparum malaria within the last 5 years.
* Prior receipt of malaria vaccine.
* Planned travel to malaria endemic areas during the study period.
* Use of drugs with known antimalarial activity within 30 days of study enrollment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin).
* Participation in other clinical trials or the intake of an investigational medicinal product within the last 90 days or planned receipt during the duration of this study
* Human Immunodeficiency Virus (HIV) infection.
* Any confirmed or suspected immunosuppressive or immunodeficient state (e.g. repeated and/or unusual infections), history of infection caused by opportunistic organisms any infection or combination of infections that suggest underlying immunodeficiency, history of meningitis, encephalitis, septic shock, life-threatening soft tissue infection, more than one pneumonia, asplenia and/or chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)).
* Use of immunoglobulins or blood products within 3 months prior to enrollment.
* Known (or signs consistent with) sickle cell anaemia, sickle cell trait, thalassemia or thalassemia trait, glucose-6-phosphate dehydrogenase deficiency.
* Pregnancy, lactation or intention to become pregnant during the study.
* Contraindications to the use of the following antimalarial medications: Atovaquone-proguanil, artemether-lumefantrine, artesunate, pyronaridine-artesunate, i.e.:

  * Known hypersensitivity to any of these drugs
  * intake of the following drugs: rifampicine, rifabutin, metoclopramide, warfarin, cumarine-derivatives, etoposide, antiretroviral drugs, imipramine, amytriptilin, clomipramin, carbamazepine, phenytoin, St. Johns wort, metoprolol, flecainide, propafenone, digoxin, dabigatran; drugs inducing QTc prolongation, drugs metabolized by CYP2D6, drugs inducing CAP3A4.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine (e.g. egg products, Kathon).
* History of clinically significant contact dermatitis.
* History of cancer within the last 5 years (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Alcohol consumption should not exceed 24 g (men) or 12 g (women)/per day
* Haemoglobin <14 g/dl (men) or <12 g/dl (women)
* Suspected or known injected drug abuse in the 5 years preceding enrollment.
* Positive for hepatitis B surface antigen (HBs-antigen).
* Seropositivity for hepatitis C virus (antibodies to HCV)
* Clinical signs or symptoms of hepatic injury (such as nausea and/or abdominal pain associated with jaundice) or known liver disease (i.e. decompensated cirrhosis, Child-Pugh stage B or C).
* Renal abnormalities
* GFR <30ml/min (glomerular filtration rate)
* Presence or past history of cardiac arrhythmia or an abnormal electrocardiogram or suspected coronary heart disease or family history for sudden cardiac death.
* Known or suspected porphyria.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* History of seizure (except uncomplicated febrile convulsion at childhood)
* Immunization with more than 3 other vaccines within four weeks.
* Electrolyte disturbance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of PfSPZ-CVac/Pyramax and MVA ME-TRAP/ChAd63 ME-TRAP | From the first administration until the last follow-up visit (Group 1: day 136, Group 2: day 82)
  Assessment of all adverse events and serious adverse events that might be related to the administration of PfSPZ-CVac/Pyramax and MVA ME-TRAP/ChAd63 ME-TRAP

SECONDARY OUTCOMES:
Assessment of protective efficacy of PfSPZ-CVac/Pyramax and of MVA ME-TRAP /ChAd63 ME-TRAP in healthy, malaria-naïve adults against homologous CHMI with PfSPZ Challenge (NF54) by DVI | From administration of CHMI (Group 1:day 113, Group 2: 59) until the last follow-up visit (Group 1: day 136, Group 2: day 82)
  Assessment of the development of parasitemias following the controlled human malaria infection (CHMI)

OTHER OUTCOMES:
Assessment of Pyramax as a drug for in vivo chemoattenuation of PfSPZ Challenge (NF54) for the PfSPZ-CVac approach | From the first administration (day 1) until the last follow-up visit (Group 1: day 136)
  Assessment of the development of parasitemias and side effects following immunization with PfSPZ-CVac and Pyramax
Assessment of the immunogenicity of each of the malaria vaccine candidates | From the first administration until the last follow-up visit (Group 1: day 136, Group 2: day 82)
  Assessment of several immungenic blood parameters and their development throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Bélard, Dr., Principal Investigator — University Hospital Tuebingen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sulyok Z, Fendel R, Eder B, Lorenz FR, Kc N, Karnahl M, Lalremruata A, Nguyen TT, Held J, Adjadi FAC, Klockenbring T, Flugge J, Woldearegai TG, Lamsfus Calle C, Ibanez J, Rodi M, Egger-Adam D, Kreidenweiss A, Kohler C, Esen M, Sulyok M, Manoj A, Richie TL, Sim BKL, Hoffman SL, Mordmuller B, Kremsner PG. Heterologous protection against malaria by a simple chemoattenuated PfSPZ vaccine regimen in a randomized trial. Nat Commun. 2021 May 4;12(1):2518. doi: 10.1038/s41467-021-22740-w. PMID 33947856